CLINICAL TRIAL: NCT03293316
Title: Using Electroencephalography (EEG) and Transcranial Current Stimulation (tCS) to Study and Modulate Cognition Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: C2-2014-033
Record Dates: First submitted 2017-09-21; First posted 2017-09-26 (Actual); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Inter-individual Variability
Keywords: Transcranial electrical stimulation; random noise;; cognitive interventions; electroencephalography;; inter-individual variability; stochastic resonance;
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Randomized Double-Blind

ARMS (3):
- Sham Transcranial Random Noise Stimulation (Sham Comparator): The sham tRNS condition involves 30 seconds of 1.5 mA tRNS, with a ramping period of 30 seconds at the onset and offset. This procedure ensures that, in both the Active and Sham conditions, participants experience the sensations associated with the onset of transcranial electrical stimulation (e.g., tingling sensation)
  Interventions: Device: Transcranial Random Noise Stimulation
- 1mA Transcranial Random Noise Stimulation (Experimental): The 1mA tRNS condition consists of 1 mA peak-to-peak (-.5 mA to .5 mA) high frequency noise (100-500 Hz), with amplitude values that are normally distributed and have a mean of zero. The stimulation is delivered for 20 minutes, with a ramping period of 30 seconds at the onset and offset.
  Interventions: Device: Transcranial Random Noise Stimulation
- 2mA Transcranial Random Noise Stimulation (Experimental): The only factor that varies for the 2mA tRNS condition is that the high frequency noise has a peak-to-peak of -1 mA to 1mA as opposed to -.5 mA to .5 mA. Again, the stimulation is delivered for 20 minutes, with a ramping period of 30 seconds at the onset and offset.
  Interventions: Device: Transcranial Random Noise Stimulation

INTERVENTIONS:
Device: Transcranial Random Noise Stimulation — The transcranial random noise stimulation was delivered using a StarStim device (Neuroelectrics®, Barcelona, Spain). The electrodes were encased in a pair of saline-soaked sponges (25 cm2 ), and were secured within a Neurolectrics EEG cap over right DLPFC (F4) and right IPL (P4), according to the 10-20 international EEG system. Other details are stated under the 'intervention arm' descriptions.
  Other Names: Starstim; Neuroelectrics

SUMMARY:
Inter-individual variability in responsiveness to interventions poses great challenges for translational neuroscience, and health care in general. The investigations sought to examine the potential for high-frequency transcranial random noise stimulation (tRNS) to modulate sustained attention in a manner that was informed by individual differences in EEG indices.

DETAILED DESCRIPTION:
Inter-individual variability in responsiveness to interventions poses great challenges for translational neuroscience, and health care in general. Reliable and cost- effective screening procedures that can identify individuals who are more likely to benefit from an intervention could have substantial real-world benefits. Here, the investigators sought to examine the potential for high-frequency transcranial random noise stimulation (tRNS) to modulate sustained attention in a manner that was informed by individual differences in a well-studied electrocortical marker, spontaneous theta/beta ratio. The investigators hypothesized that individuals with relatively high theta/beta ratios, putatively reflecting suboptimal cortical arousal, would be more likely to benefit from the gains in cortical excitability afforded by tRNS. Seventy-two young healthy adults were administered 1mA, 2mA and sham tRNS in a double-blind, randomised, cross-over manner, while they performed a continuous monitoring paradigm. Electroencephalography was acquired before and after each stimulation condition.

This approach may constitute a feasible means of using individual differences in neurophysiology to inform predictions about outcomes from targeted cognitive interventions.

ELIGIBILITY:
Inclusion criteria:

- Aged 18-35 years

Exclusion criteria:

* Left-handedness
* Visual impairment
* History of fainting,
* History of neurological or psychiatric illness,
* Neurological insult
* Drug or alcohol abuse
* Reporting current use of anti- psychotic or anti-depressant medications

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Electroencephalography | 4 minutes
  Voltage readings from the scalp

SECONDARY OUTCOMES:
Sustained Attention performance | 20 minutes
  Sustained Attention performance was defined as response time variability on a continuous monitoring paradigm